CLINICAL TRIAL: NCT03797430
Title: Determination of Normal Values for the Star Excursion Balance Test(SEBT) in National or International Handball Young Women Players
Brief Title: Determination of Normal Values for the Star Excursion Balance Test (SEBT) in Handball Players
Acronym: SEBTHAND
Status: Withdrawn | Type: Observational
Why Stopped: NO PARTICIPANTS ENROLLED
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: SEBTHAND ( 29BRC18.0254)
Record Dates: First submitted 2019-01-02; First posted 2019-01-09 (Actual); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Handball Players
Keywords: hand ball; evaluation; risk of injury; women

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
the aim of this study is to determine normal values for SEBT in young national or international handball women players for determining specific level for SEBT to predict risk of injury

ELIGIBILITY:
Inclusion Criteria:

* women
* age from 14 to 18 years old
* national or international level for handball

Exclusion Criteria:

* no french language
* players who don't understand the instructions to perform the test
* Refusal to perform the test

Ages: 14 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — handball women players
Study Population: national or international hanball women players, aged from 14 to 18 years old
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-01-02 (Estimated); Primary Completion 2020-01-02 (Estimated); Study Completion 2020-01-02 (Estimated)

PRIMARY OUTCOMES:
determination of normal values for SEBT | one day
  star excursion balance test : it is a functionnal test for predicting the risk of injury

CONTACTS AND LOCATIONS:
Overall Officials: Marc BEAUMONT, PhD, Principal Investigator — CHU Brest